CLINICAL TRIAL: NCT01782417
Title: Pilot Testing a Patient and Provider Intervention for Managing Osteoarthritis in Hispanic Adults.
Acronym: PRIMO-Latino
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00022836_1
Record Dates: First submitted 2013-01-31; First posted 2013-02-01 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-06

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis; Hispanic; behavior; intervention; Spanish
MeSH Terms: conditions — Osteoarthritis; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient and provider intervention (Other): participants will receive a patient and provider intervention
  Interventions: Behavioral: patient and provider intervention

INTERVENTIONS:
Behavioral: patient and provider intervention — Patients receive a 12-month intervention consisting of monthly phone calls focusing on exercise, weight management, and cognitive behavioral pain management; primary care providers receive patient-specific osteoarthritis information and treatment recommendations at the point of clinical care.

SUMMARY:
Hispanics are affected by arthritis at a slightly lower age-adjusted rate compared to non-Hispanic whites and African Americans. However, compared to other groups, Hispanics have a higher prevalence of arthritis-attributed activity limitations (primarily related to OA), are less likely to receive hip replacement independent of health care access, and are less likely to receive knee replacement. The study is conducted to develop and test a telephone delivered intervention for the management of OA in Hispanic adults. This study is conducted as a minority supplement to the Patient and Provider Interventions for Managing Osteoarthritis in Primary Care (PRIMO) NCT01435109 and Pro00022836.

DETAILED DESCRIPTION:
Arthritis affects approximately 50 million adults in the United States (US), making it one of the most common causes of disability in this county. In addition, is associated with significant physical activity limitations, increased prevalence of obesity, decreased health related quality of life, and increased health care costs. Hispanics are affected by arthritis at a slightly lower age-adjusted rate compared to non-Hispanic whites and African Americans. However, compared to other groups, Hispanics have a higher prevalence of arthritis-attributed activity limitations (primarily related to OA), are less likely to receive hip replacement independent of health care access, and are less likely to receive knee replacement. In addition, there have been very few interventions to improve either medical or behavioral aspects of OA treatment recommendations among the Hispanic population. The study will developed and test a culturally appropriate Spanish educational materials and telephone scripts for the patient- and provider-based interventions and will test the patient and provider intervention in a group of Adult Hispanics with OA.

ELIGIBILITY:
Inclusion Criteria:

* Radiographic evidence of hip OA and/or radiographic evidence of or meets clinical criteria for knee OA
* Current joint (hip and/or knee) symptoms
* BMI >= 25
* Physically inactive
* Spanish speakers

Exclusion Criteria:

* Diagnosis of rheumatoid arthritis, fibromyalgia, or other systemic rheumatic disease
* Diagnosis of a motor neuron disease, Parkinson's disease, multiple sclerosis, or Paget's disease
* Diagnosis of metastatic cancer
* Hospitalized for a stroke, myocardial infarction or coronary artery revascularization in the past 3 months
* On waiting list for or planning arthroplasty
* Total joint replacement (hip or knee) surgery, other hip or knee surgery, meniscus tear (verified by MRI), or (anterior cruciate ligament) ACL tear in the past 6 months
* History of gout in hip or knee
* Quadriplegia or paraplegia
* Active diagnosis of psychosis or serious personality disorder
* Diagnosis of dementia or other memory loss condition
* Current, uncontrolled substance abuse disorder
* Severly impaired speech or hearing (patients must be able to respond to phone calls)
* No access to a telephone
* Resident in nursing home
* Serious / terminal illness as indicated by referral to hospice or palliative care
* For females: currently pregnant or planning to become pregnant
* Participating in another OA intervention of other lifestyle change study
* Other self-reported medical problem that would prohibit participation in the study
* Other health condition or personal issue judged by a study team member or primary care physician to make the patient inappropriate for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in Self-reported pain, stiffness and function. | baseline, 6 months and 12 months.
  Measured by the validated Spanish version of the Western Ontario and McMasters Universities Osteoarthritis Index (WOMAC).

SECONDARY OUTCOMES:
Change in Physical function | Baseline and 12 months
  Short Physical Performance Test Protocol
Change in Depressive symptoms | Baseline and 12 months
  Measured with the Spanish version of the Patient Health Questionnaire (PHQ-8).
Change in weight | Baseline and 12 months
  measured on a standard scale
Participants perception of the intervention | 12 months
  Semi structured interviews

CONTACTS AND LOCATIONS:
Overall Officials: Kelli Allen, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Corsino L, Coffman CJ, Stanwyck C, Oddone EZ, Bosworth HB, Chatterjee R, Jeffreys AS, Dolor RJ, Allen KD. A feasibility study to develop and test a Spanish patient and provider intervention for managing osteoarthritis in Hispanic/Latino adults (PRIMO-Latino). Pilot Feasibility Stud. 2018 Jul 4;4:89. doi: 10.1186/s40814-018-0280-x. eCollection 2018. PMID 29997898